CLINICAL TRIAL: NCT05789368
Title: Efficacy Testing of VeCollal Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 22-112-A
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Skin Condition
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo sachet (Placebo Comparator): consume 1 sachet per day
  Interventions: Dietary Supplement: Placebo sachet
- VeCollal sachet (Experimental): consume 1 sachet per day
  Interventions: Dietary Supplement: VeCollal sachet
- Collagen sachet (Active Comparator): consume 1 sachet per day
  Interventions: Dietary Supplement: Collagen sachet

INTERVENTIONS:
Dietary Supplement: Placebo sachet — consume 1 sachet per day
  Arms: Placebo sachet
Dietary Supplement: VeCollal sachet — consume 1 sachet per day
  Arms: VeCollal sachet
Dietary Supplement: Collagen sachet — consume 1 sachet per day
  Arms: Collagen sachet

SUMMARY:
To assess VeCollal formula on skin condition improvement

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged above 20 years old

Exclusion Criteria:

* Subject who is not willing to participate in this study.
* Patients with diseases of the skin, liver, kidney.
* Subjects who have known cosmetic, drug or food allergies, difficulty in digestive tract absorption or disorder.
* Female who is pregnant or nursing or planning to become pregnant during the course of the study.
* Received facial laser therapy, chemical peeling or UV overexposure (> 3 hr/week) in the past 4 weeks.
* Constant drug use
* Students who are currently taking courses taught by the principal investigator of this trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
The change of skin collagen density | Change from Baseline skin collagen density at 8 weeks
  DermaLab® Series SkinLab Combo was utilized to measure skin pores. Units: arbitrary units
The change of skin wrinkles | Change from Baseline skin wrinkles at 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin wrinkles. Units: arbitrary units
The change of skin texture | Change from Baseline skin texture at 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin texture. Units: arbitrary units
The change of skin elasticity | Change from Baseline skin elasticity at 8 weeks
  SoftPlus was utilized to measure skin elasticity. Units: arbitrary units

SECONDARY OUTCOMES:
The change of skin melanin index | Change from Baseline skin melanin index at 8 weeks
  Mexameter® MX18 was utilized to measure skin melanin index. Units: arbitrary units
The change of skin L* value | Change from Baseline skin L* value at 8 weeks
  Chroma Meter MM500 was utilized to measure skin L* value. Units: arbitrary units, 0-100
The change of skin erythema index | Change from Baseline skin erythema index at 8 weeks
  Mexameter® MX18 was utilized to measure skin erythema index. Units: arbitrary units
The change of skin moisture | Change from Baseline skin moisture index at 8 weeks
  Corneometer® CM825 was utilized to measure skin moisture. Units: arbitrary Corneometer® units 0-120
The change of transepidermal water loss (TEWL) | Change from Baseline skin TEWL at 8 weeks
  Tewameter® TM 300 was utilized to measure TEWL. Units: g/hm²
The change of skin pores | Change from Baseline skin pores at 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin pores. Units: arbitrary units

OTHER OUTCOMES:
The change of liver function biomarkers (AST, ALT) of blood | Change from Baseline liver function biomarkers at 8 weeks
  Fasting venous blood was sampled to measure liver function biomarkers
The change of renal function biomarkers (creatinine, BUN) of blood | Change from Baseline renal function biomarkers at 8 weeks
  Fasting venous blood was sampled to measure renal function biomarkers
The change of fasting blood glucose | Change from Baseline blood glucose at 8 weeks
  Fasting venous blood was sampled to measure blood glucose
The change of blood lipid profiles (total cholesterol, triglyceride) | Change from Baseline blood lipid profiles at 8 weeks
  Fasting venous blood was sampled to measure blood lipid profiles
The change of self-assessment skin condition | Change from Baseline skin condition at 8 weeks
  A self-assessment questionnaire was collected to evaluate skin condition

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hua Liang, Principal Investigator — Chia Nan University of Pharmacy ＆ Science
Locations (1):
- Chia Nan University of Pharmacy ＆ Science, Tainan, Taiwan